CLINICAL TRIAL: NCT01320540
Title: 4R (Right Information and Right Care to the Right Patient at the Right Time) for Guideline Indicated BRCA Genetic Assessment of Breast Center Patients
Brief Title: 4R for Guideline Indicated BRCA Testing of Breast Center Patients
Acronym: 4R
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Melissa Simon, Associate Professor, Northwestern University
Other Study IDs: STU00041300
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Newly Diagnosed Carcinoma of Breast; Genetic Predisposition to Disease
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Breast Center Patients: Patients newly diagnosed with breast cancer who did or did not have genetic testing (retrospectively and prospectively).
- Staff from the Lynn Sage Comprehensive Breast Cancer Center: Members of the Northwestern staff to include but not limited the Lynn Sage Comprehensive Breast Cancer Center and/or Breast Cancer Genetics Program provider staff (including physicians, nurses, schedulers, physician assistants and/or genetic counselors).

SUMMARY:
Currently, many breast center patients with a positive family history receive information about BRCA testing after breast cancer diagnosis, typically after definitive breast surgery or at a time point that does not allow them to use testing results in making their surgical decision. Diagnostics, decisions and interventions are often out of sequence, resulting in test information not available in time for decisions. Tests are often repeated. Decisions and interventions are delayed, are not understood by breast cancer patients or proceed without the test information, resulting in suboptimal care and resource waste (Donaldson MS. 2005, Katz SJ 2007, IOM 2001).

In this study, BRCA testing information will be delivered to patients at the point of breast imaging. For patients that are diagnosed with breast cancer, this provides ample time to use the test results in making their surgical decision, if they elect to be tested. The investigators will work with health care providers to insure family history data are collected at the breast imaging visit, develop a standardized BRCA patient education handout, enlist health care providers to insure the information is delivered to the appropriate patient population, and coordinate scheduling with genetic counseling services to insure patients are promptly seen.

The investigators hypothesis is that an intervention of providing patients indicated for genetic/familial risk with timely information and opportunity to access genetic counseling during breast imaging will shift BRCA testing to before definitive breast cancer surgery, for patients with a breast cancer diagnosis, and could impact surgical decisions. The investigators will identify barriers to this intervention from the perspective of patients, physicians, nurses, and genetic counselors. The investigators will then adjust the intervention to overcome the barriers and will test the intervention at the point where genetic/familial risk assessment based on NCCN guidelines is (or should be) conducted at breast imaging. If indicated, patients will be provided information and will be referred to genetic counseling to consider BRCA tests.

DETAILED DESCRIPTION:
This study is expected to involve a total of 2,101 individuals: 89 (83 for testing the intervention and 6 who participated in interviews like Northwestern staff participants) breast cancer patients, 12 Northwestern staff,and 2,000 women who consented and participated in the genetics assessment screening survey using the tool, with a sub-cohort of 300 that may benefit from genetic assessment and/or testing based on the screening tool results.

All subjects will be assigned a unique study number to minimize the risk of a breach of confidentiality. This is the only anticipated risk to subjects participating in this study utilizing retrospective and prospective chart reviews and interviews.

TESTING THE INTERVENTION

Investigators will collect retrospective data for 83 breast cancer patients diagnosed who underwent BRCA testing and definitive breast cancer surgery at Northwestern between 07/01/2008 to 06/30/2010. This baseline information detailed on the Data Collection Form will be collected using EDW and NMFF and NMH medical record systems.

The intervention involves radiologists who convey pathology results to patients with suspected breast cancers. At the time the patient with a familial/ genetic risk is informed of a positive test result for breast cancer, the radiologist will provide information about genetic counseling and offer to send an educational handout via e-mail or regular mail. This intervention will be conducted with newly diagnosed breast cancer patients between 03/01/2011and 05/31/2012.

Investigators will prospectively collect data on these 83 breast cancer patients who are diagnosed, received BRCA testing, and had definitive surgery at Northwestern during the time of the intervention, 03/01/2011 and 05/31/2012. The EDW and NMFF and NMH medical record systems will be used to collect this information.

Because the intervention and retrospective and prospective chart reviews pose minimal risk to the subjects and locating the patients or having access to the patients would be time and cost prohibitive, a waiver of consent and HIPAA is requested.

ASSESS IMPACT OF THE INTERVENTION

Study investigators will conduct interviews with a total of 6 breast cancer patients and 12 Northwestern staff to determine if the intervention improved the care process. Written consent will be obtained from all interview participants. Participants will have the option of being audiotaped. Audiotaping is not required.

* Prior to the intervention, investigators will interview 6 breast cancer patients and 12 Northwestern staff to find out about the current care process and opinions/feedback on proposed intervention.
* Following the intervention, 6 patients and 12 staff will be interviewed using the same questions and format. It is acceptable that the individuals participating in the post-intervention interview are not the same as those participating in the pre-intervention interview.

INTERVENTION TEST/INTERVENTION IMPLEMENTATION

The intervention will be tested with women age 18 and older who have a history of genetic/familial risk and patients at the Lynn Sage Comprehensive Breast Center between March 1, 2013 and February 28, 2014. There will be no follow up on these patients after March 31, 2014..

1. Select breast center patients who consent to participate in this study will take a basic familial/genetic risk survey that follows NCCN guidelines (up to 2,000 patients will be consented into this study, with a sub-cohort of up to 300 who are identified to have a familial / genetic risk for breast cancer. If no risk is identified, the patient is not specifically informed of genetic counseling.
2. For study consented breast center patients with familial / genetic risk, the cancer genetics program will provide information about genetic counseling. The research staff will track those patients who receive information about genetic counseling.

ELIGIBILITY:
Inclusion Criteria:

Retrospective chart review of 83 breast cancer patients:

* Female
* Age 18 and older
* Diagnosed with invasive breast cancer at Northwestern between 07/01/2008 and 06/30/2010

Prospective chart review of 83 patients:

* Female
* Age 18 and older
* Diagnosed with invasive breast cancer at Northwestern between 03/01/2011 and 05/31/2012

For patient interviews:

* Female
* Age 18 and older
* Are not inpatients
* Patients seen at the Lynn Sage Comprehensive Breast Center

For staff interviews:

Members of the Northwestern staff to include but not limited the Lynn Sage Comprehensive Breast Cancer Center and/or Breast Cancer Genetics Program provider staff (including physicians, nurses, schedulers, physician assistants and/or genetic counselors)

Exclusion Criteria:

* Under 18 years of age

To test the intervention, patients seen at the breast center:

* Are female
* Are age 18 and older
* Are not institutionalized
* Are being seen at the Lynn Sage Comprehensive Breast Center
* Have a positive family history per NCCN guidelines on genetic/familial high risk assessment for breast and ovarian cancer

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women newly diagnosed with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The timing of genetic testing in regards to what kind of surgery was performed | 36 months
  To test an intervention for breast cancer patients with familial/genetic risk by obtaining data on 83 women with breast cancer who were tested before the intervention was implemented and comparing their outcomes to 83 women with breast cancer who were treated after the intervention was implemented. The primary endpoint is the timing of BRCA testing relative to (before or after) definitive breast cancer surgery and the surgical decision (lumpectomy, mastectomy, bi-lateral mastectomy).
The timing of genetic testing in regards to what kind of surgery was performed | 12 months
  To test an intervention for breast center patients with familial/genetic risk by obtaining data on 2,000 women who consented and participated in the genetics assessment screening survey, with a sub-cohort of 300 that may benefit from genetic assessment and/or testing based on the screening tool results.

SECONDARY OUTCOMES:
Impact of the intervention | 36 months
  To assess the care process impact of the intervention on patients and provider staff through pre and post intervention interviews. The process impact will be assessed by comparing the questionnaires from the pre and post intervention interviews in 6 patients and 12 providers.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Simon, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States